CLINICAL TRIAL: NCT02818010
Title: Impact of Physical Activity on Patients With Chronic Kidney Disease Not Receiving Dialysis Followed in the TIRCEL Network. An Exposed / Unexposed Study (PHYSALYS)
Acronym: PHYSALYS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50806
Record Dates: First submitted 2016-06-21; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: physical activity; chronic kidney disease; nephrology; stage 3; stage 4; stage 5
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- exposed = patient practicing physical activity: The practice of physical activity is measured by the GPAQ 2 questionnaire (Global Physical Activity Questionnaire)
  A patient is defined as practicing physical activity (exposed) when he meets one of the conditions following:
  * At least 20 minutes of vigorous-intensity physical activity for at least 3 days per week
  * At least 30 minutes of moderate-intensity physical activity or walking daily for at least 5 days per week
  * At least 5 days of walking and moderate- or vigorous-intensity physical activity achieving at least 600 MET-minutes per week.
  The Metabolic equivalents (MET) is the ratio of metabolic rate during activity physical and metabolic rate at rest. One MET corresponds to the energy spent by a person sitting still and is equivalent to a consumption of 1 kcal / kg / hour. It is estimated that a moderately active person has an energetic cost four times higher, and a very active person eight times higher than the energy cost of a person sitting without move.
  Interventions: Other: Global Physical Activity Questionnaire
- unexposed = patient not practicing physical activity: The practice of physical activity is measured by the GPAQ 2 questionnaire(Global Physical Activity Questionnaire)
  A patient is defined as unexposed if he does not fulfill any of these conditions :
  * At least 20 minutes of vigorous-intensity physical activity for at least 3 days per week
  * At least 30 minutes of moderate-intensity physical activity or walking daily for at least 5 days per week
  * At least 5 days of walking and moderate- or vigorous-intensity physical activity achieving at least 600 MET-minutes per week.
  The Metabolic equivalents (MET) is the ratio of metabolic rate during activity physical and metabolic rate at rest. One MET corresponds to the energy spent by a person sitting still and is equivalent to a consumption of 1 kcal / kg / hour. It is estimated that a moderately active person has an energetic cost four times higher, and a very active person eight times higher than the energy cost of a person sitting without move.
  Interventions: Other: Global Physical Activity Questionnaire

INTERVENTIONS:
Other: Global Physical Activity Questionnaire — The practice of physical activity is measured by the GPAQ 2 questionnaire (Global Physical Activity Questionnaire) developed by the World Health Organization.

SUMMARY:
PHYSALYS is an observational multicenter study. It's an analytical study comparing 2 groups: patients exposed to physical activity and unexposed. The main objective of the study is to compare the evolution of glomerular filtration rate at inclusion and 12 months later between patients practicing physical activity and patients not practicing. If necessary, the renal disease-related complications, which are not influenced by physical activity: (type of kidney disease, age and tobacco), would be taken into account. TIRCEL patients with chronic kidney disease (CKD) at stages 3, 4 or 5 can be included in the study. Their serum creatinine data, 12 months prior to inclusion, is collected retrospectively. Patients are followed in the trial during 12 months. To evaluate physical activity, patients respond to Global Physical Activity Questionnaire 2 (GPAQ2) at inclusion and 12 months later. During this 12 months period, the same biological data are collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Members of TIRCEL (Traitement de l'Insuffisance Chronique en rhônE-aLpes) network for over a year and having at least two measurements of glomerular filtration rate with an interval of 9 to 12 months between the first and the last measurement
* Patients in stages 3, 4 or 5 of CKD
* No dialysis CKD patients
* Non transplanted CKD patients
* Patients seeing nephrologist
* Patients agreeing to be contacted for a phone call half an hour
* Adults patients (> 18 years)
* Patients not living in institution
* Patients being able to answer a questionnaire

Exclusion Criteria:

* Patients followed in the TIRCEL (Traitement de l'Insuffisance Chronique en rhônE-aLpes) network for less than one year or having less than 2 measurements of glomerular filtration rate with an interval of least 9 months or over 12 months between the first and the last measurement
* Patients in stages 1 or 2 of CKD
* CKD patients receiving dialysis
* Transplanted CKD patients
* Patients not seeing nephrologist
* Patients refusing to be contacted for a phone call half an hour
* Patients < 18 years
* Patients living in institution
* Patients unable to answer a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients ( ≥ 18 years); members of TIRCEL network for over a year and having at least two measures of glomerular filtration rate with an interval of at least 9 to 12 months between the first and the last measurement; in CKD stage 3,4 or 5; not on dialysis and not transplanted, making a visit to their nephrologist; agreeing to be contacted at home for a phone call half an hour; not living in institution and being able to answer a questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2012-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change of the Glomerular Filtration Rate (GFR) | Month 0, Month 12
  The Glomerular Filtration Rate (GFR) annual slope between inclusion (M0) and 12 months (M12) after inclusion in exposed and unexposed groups.